CLINICAL TRIAL: NCT00508170
Title: Sexual Behavior in Oropharyngeal Patients Versus Head and Neck Cancer Patients, With or Without HPV Infection
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0519
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Cancer; Oropharyngeal Cancer; Human Papillomavirus Infection
Keywords: Head and Neck Cancer; Human Papillomavirus Infection; Oropharyngeal Patients; Sexual Behavior; Questionnaire
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Papillomavirus Infections; Sexual Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Oropharyngeal Cancer
  Interventions: Behavioral: Questionnaire
- Patients with Non-Oropharyngeal Cancer
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — The questionnaire contains 23 questions and is estimated to take approximately 10 minutes to complete.

SUMMARY:
Primary Objectives:

1. To determine whether high-risk sexual behaviors are more common in patients with oropharyngeal cancer than in patients with head and neck cancers of other sub-sites.
2. To determine if high-risk sexual behaviors are more common in patients with HPV (human papillomavirus) associated head and neck cancer than those without evidence of HPV-16 infection.

DETAILED DESCRIPTION:
Squamous cell cancer of the head and neck (SCCHN) is believed to be caused by the long-term exposure of the mucous membrane on the inside of the mouth to different types of cancer-causing agents. This results in changes in the mouth, which can lead to the development of cancer.

Infection with HPV-16 has been linked with SCCHN. Half of all cancers of the oropharynx (the middle part of the throat including the soft palate, base of the tongue, and tonsils) are caused by HPV-16. HPV-16 is normally sexually transmitted, and is the cause of cervical cancer in women. By finding out if the virus is also sexually transmitted to the oropharynx, doctors may be able to educate patients about risk factors for developing cancer in this region. Eventually, doctors may be able to vaccinate people who are at risk for getting this virus.

You have received this questionnaire because you gave researchers your verbal consent for the mail-out. Along with the questionnaire, included are 2 self-addressed stamped envelopes for you to return the questionnaire and consent separately.

If you agree to take part in this study, you will complete the questionnaire about your sexual history such as specific sexual practices and number of partners, exposure to HPV and other viruses, and any relevant medical history. This questionnaire should take about 10 minutes to complete. The questionnaire will be given a study code number so that your name or M. D. Anderson patient ID number will not appear on the questionnaire.

Once you have finished the questionnaire, for added privacy and confidentiality, you should place the signed consent form in 1 self-addressed stamped envelope (SASE) and the completed questionnaire into the other self-addressed stamped envelope (SASE) that has been provided. Please mail both envelopes back within 15 days of receiving the questionnaire.

Once you have completed the questionnaire, your participation in this study is over.

This is an investigational study. About 1,267 patients will be enrolled in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosed squamous cell carcinoma of the head and neck that participated in the molecular epidemiology study LAB00-062 of head and neck cancer between 1995 and 2005.
2. Head and Neck cancer participants of LAB00-062 that are still alive.
3. Head and Neck cancer participants of LAB00-062 that have known mailing addresses in the U.S.A.
4. Patients must be 18 years and older.
5. Patients will have completed their primary treatment but may be undergoing treatment for a second primary or recurrent disease.
6. Ability to read, write, and speak Spanish or English.

Exclusion Criteria:

n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed squamous cell carcinoma of the head and neck that participated in the molecular epidemiology study LAB00-062 of head and neck cancer between 1995 and 2005.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Number of Responders with High-risk Sexual Behaviors | 1 month for mailing and return of questionnaires
  Written self-administered questionnaire responses analyzed to determine whether patients with oropharyngeal cancer have history of high-risk sexual behavior (defined as 15 or more lifetime sexual partners) greater than that of patients with tumors of other sites of head and neck

CONTACTS AND LOCATIONS:
Overall Officials: Erich Sturgis, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://mdanderson.org